CLINICAL TRIAL: NCT00467740
Title: Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study to Assess the Efficacy (Bronchodilation) and Safety of 4 Weeks of Treatment of Orally Inhaled BI 1744 CL (4 Doses) Delivered by the Respimat® Inhaler in Patients With Asthma
Brief Title: Efficacy and Safety of 4 Weeks of Treatment With Inhaled BI 1744 CL in Patients With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1222.6; EUDRACT 2006-004829-29
Record Dates: First submitted 2007-04-30; First posted 2007-05-01 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — olodaterol

INTERVENTIONS:
Drug: BI 1744 CL

SUMMARY:
The primary objective of this study is to determine the optimum dose(s) of BI 1744 CL inhalation solution delivered by the Respimat® inhaler for four weeks in patients with asthma. The selection of the optimum dose(s) will be based on bronchodilator efficacy (how well it helps your breathing), safety evaluations and pharmacokinetic evaluations (the amount of the medication found in your blood).

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent consistent with ICH-GCP guidelines prior to participation in the trial, which includes medication washout and restrictions
2. Male or female patients, 18 years of age or older
3. Diagnosis of asthma (GINA)
4. Pre-bronchodilator FEV1 greater than or equal to 60% predicted and <90% predicted (ECSC);
5. Increase in FEV1 greater than or equal to 12% and 200 ml 15 minutes after 400µg salbutamol (albuterol) at Visit 1
6. Patient must have been taking Inhaled Corticosteroids for at least 12 weeks prior to screening, and must have been receiving a stable low/moderate dose for at least 6 weeks prior to screening.
7. Patients must be able to perform technically acceptable pulmonary function tests and PEF measurements, and must be able to maintain records (Patient Daily e-Diary) during the study period as required in the protocol
8. Patients must be able to inhale medication in a competent manner from the Respimat® inhaler and from a metered dose inhaler (MDI).

Exclusion Criteria:

1. Patients with a smoking history of more than 10 pack years
2. Patients with any of the following conditions: a diagnosis of thyrotoxicosis, a diagnosis of paroxysmal tachycardia (>100 beats per minute), a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms), a history of additional risk factors for Torsade de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
3. Patients with any of the following conditions: a history of myocardial infarction within 1 year of screening visit (Visit 1), a diagnosis of clinically relevant cardiac arrhythmia, a history of cor pulmonale, known active tuberculosis, a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with treated basal cell carcinoma are allowed), a history of life-threatening pulmonary obstruction, a history of cystic fibrosis, clinically evident bronchiectasis, a history of significant alcohol or drug abuse
4. Patients who have undergone thoracotomy with pulmonary resection
5. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Visit (Visit 1)
6. Pregnant or nursing women
7. Women of childbearing potential not using a highly effective method of birth control. Female patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation, or post-menopausal for at least 2 years
8. Patients who have previously been randomized in this study or are currently participating in another study
9. Patients who are unable to comply with pulmonary medication restrictions prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2007-05; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (37):
- United States (10):
  - 1222.6.064 Arthur F. Gelb Medical Corporation, Lakewood, Lakewood, California
  - 1222.6.062 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1222.6.066 Allergy & Asthma Medical Group and Rsrch Ctr, APC, San Diego, California
  - 1222.6.069 Allergy Associates Medical Group, San Diego, California
  - 1222.6.068 National Jewish Medical Center, Denver, Colorado
  - 1222.6.073 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1222.6.067 Northeast Medical Research Associates, Inc, North Darthmouth, Massachusetts
  - 1222.6.061 Center for Human Genomics, Winston-Salem, North Carolina
  - 1222.6.072 Boehringer Ingelheim Investigational Site, Kileen, Texas
  - 1222.6.071 Pulmonary Consultants, Tacoma, Washington
- Canada (14):
  - 1222.6.017 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1222.6.006 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1222.6.012 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1222.6.016 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1222.6.011 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1222.6.003 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 1222.6.013 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1222.6.005 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1222.6.009 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1222.6.008 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1222.6.015 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1222.6.007 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
  - 1222.6.002 Boehringer Ingelheim Investigational Site, Ste-Foy, Quebec
  - 1222.6.004 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- France (7):
  - 1222.6.3303A Boehringer Ingelheim Investigational Site, Béthune
  - 1222.6.3308A Boehringer Ingelheim Investigational Site, Briançon
  - 1222.6.3302A Boehringer Ingelheim Investigational Site, Grenoble
  - 1222.6.3306A Boehringer Ingelheim Investigational Site, Lille
  - 1222.6.3301A Boehringer Ingelheim Investigational Site, Montpellier
  - 1222.6.3304A Boehringer Ingelheim Investigational Site, Nîmes
  - 1222.6.3305A Boehringer Ingelheim Investigational Site, Saint-Pierre Cedex - La Réunion
- Germany (6):
  - 1222.6.031 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.6.034 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.6.037 Boehringer Ingelheim Investigational Site, Gauting
  - 1222.6.038 Boehringer Ingelheim Investigational Site, Hamburg
  - 1222.6.032 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 1222.6.036 Boehringer Ingelheim Investigational Site, Wiesloch

REFERENCES:
- [Derived] O'Byrne PM, D'Urzo T, Beck E, Flezar M, Gahlemann M, Hart L, Blahova Z, Toorawa R, Beeh KM. Dose-finding evaluation of once-daily treatment with olodaterol, a novel long-acting beta2-agonist, in patients with asthma: results of a parallel-group study and a crossover study. Respir Res. 2015 Aug 18;16(1):97. doi: 10.1186/s12931-015-0249-8. PMID 26283085

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler.
- Olo 2 mcg qd: Olodaterol 2 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 5 mcg qd: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 20 mcg qd: Olodaterol 20 mcg qd (morning) delivered by the Respimat Inhaler.
Period: Overall Study
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Started | 54 | 61 | 60 | 60 | 61
Completed | 53 | 58 | 58 | 59 | 61
Not Completed | 1 | 3 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Total
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.59 (14.11) | 45.36 (15.12) | 46.17 (12.96) | 46.25 (14.45) | 44.62 (12.95) | 45.23 (13.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 39 | 30 | 34 | 33 | 170
  Male | 20 | 22 | 30 | 26 | 28 | 126

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1 Response After 4 Weeks
Description: Response was defined as change from baseline. Baseline trough FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed just prior to first dose of randomized treatment. Trough FEV1 is defined as the FEV1 performed at -10 mins prior to study drug inhalation at the end of the dosing interval.
Time Frame: Baseline and 4 weeks
Population: Full analysis set (FAS) is defined as all randomized patients who received at least one dose of treatment and had baseline data for at least one endpoint.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 53 | 61 | 59 | 60 | 61
Liter | 0.004 (0.034) | 0.083 (0.032) | 0.090 (0.032) | 0.080 (0.032) | 0.150 (0.032)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0754, Mixed Models Analysis; Mixed effect model with terms baseline, treatment, test day, baseline-by-test-day, treatment-by-test-day, and center as random effect; Mean Difference (Final Values) = 0.080, 95% CI [-0.008 to 0.167], Standard Error of Mean 0.045 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0571, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 0.086, 95% CI [-0.003 to 0.174], Standard Error of Mean 0.045 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0906, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.076, 95% CI [-0.012 to 0.164], Standard Error of Mean 0.045 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.147, 95% CI [0.059 to 0.234], Standard Error of Mean 0.044 — Olo 20 mcg qd minus Placebo

2. Secondary Outcome: Weekly Mean Pre-dose Morning PEFR After 4 Weeks
Description: Response was defined as change from baseline. Baseline peak expiratory flow response (PEFR) was defined as the mean of the morning PEFR measurements obtained during the week just prior to first dose of randomized treatment.
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter/minute
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 59 | 61
Liter/minute | 368.18 (5.713) | 384.42 (5.377) | 396.06 (5.419) | 404.26 (5.465) | 411.13 (5.377)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0393, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 16.238, 95% CI [0.801 to 31.675], Standard Error of Mean 7.843 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 27.878, 95% CI [12.379 to 43.378], Standard Error of Mean 7.875 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 36.072, 95% CI [20.512 to 51.633], Standard Error of Mean 7.906 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 42.943, 95% CI [27.498 to 58.389], Standard Error of Mean 7.848 — Olo 20 mcg qd minus Placebo

3. Secondary Outcome: Trough FEV1 Response After 1 Week
Description: as for outcome 1
Time Frame: Baseline and 1 week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 53 | 61 | 59 | 60 | 61
Liter | -0.007 (0.033) | 0.060 (0.031) | 0.094 (0.032) | 0.106 (0.031) | 0.166 (0.031)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.1264, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.067, 95% CI [-0.019 to 0.154], Standard Error of Mean 0.044 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0232, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.101, 95% CI [0.014 to 0.188], Standard Error of Mean 0.044 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0106, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.114, 95% CI [0.027 to 0.200], Standard Error of Mean 0.044 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.173, 95% CI [0.087 to 0.260], Standard Error of Mean 0.044 — Olo 20 mcg qd minus Placebo

4. Secondary Outcome: Trough FEV1 Response After 2 Weeks
Description: as for outcome 1
Time Frame: Baseline and 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 53 | 61 | 59 | 60 | 61
Liter | -0.009 (0.036) | 0.094 (0.034) | 0.080 (0.034) | 0.034 (0.034) | 0.131 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0329, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.103, 95% CI [0.008 to 0.198], Standard Error of Mean 0.048 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0666, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.089, 95% CI [-0.006 to 0.184], Standard Error of Mean 0.048 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.3738, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.043, 95% CI [-0.052 to 0.137], Standard Error of Mean 0.048 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0037, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.140, 95% CI [0.046 to 0.234], Standard Error of Mean 0.048 — Olo 20 mcg qd minus Placebo

5. Secondary Outcome: Trough FVC Response After 1 Week
Description: Response was defined as change from baseline. Baseline trough FVC was defined as the mean of the -1 hour and -10 minute measurements performed just prior to first dose of randomized treatment. Trough FVC is defined as the FVC performed at -10 mins prior to study drug inhalation at the end of the dosing interval.
Time Frame: Baseline and 1 week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 53 | 61 | 59 | 60 | 61
Liter | 0.001 (0.036) | 0.053 (0.034) | 0.044 (0.034) | 0.070 (0.034) | 0.131 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.2646, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.051, 95% CI [-0.039 to 0.142], Standard Error of Mean 0.046 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.3527, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 0.043, 95% CI [-0.048 to 0.135], Standard Error of Mean 0.046 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1369, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.069, 95% CI [-0.022 to 0.160], Standard Error of Mean 0.046 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0051, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.130, 95% CI [0.039 to 0.221], Standard Error of Mean 0.046 — Olo 20 mcg qd minus Placebo

6. Secondary Outcome: Trough FVC Response After 2 Weeks
Description: as for outcome 5
Time Frame: Baseline and 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 53 | 61 | 59 | 60 | 61
Liter | -0.029 (0.041) | 0.098 (0.039) | 0.069 (0.039) | -0.002 (0.038) | 0.100 (0.038)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0170, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.127, 95% CI [0.023 to 0.232], Standard Error of Mean 0.053 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0646, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.099, 95% CI [-0.006 to 0.204], Standard Error of Mean 0.053 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.6020, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.028, 95% CI [-0.077 to 0.132], Standard Error of Mean 0.053 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0147, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.130, 95% CI [0.026 to 0.233], Standard Error of Mean 0.053 — Olo 20 mcg qd minus Placebo

7. Secondary Outcome: Trough FVC Response After 4 Weeks
Description: as for outcome 5
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 53 | 61 | 59 | 60 | 61
Liter | 0.018 (0.041) | 0.055 (0.039) | 0.076 (0.039) | 0.042 (0.039) | 0.166 (0.038)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.4902, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.037, 95% CI [-0.068 to 0.142], Standard Error of Mean 0.053 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.2832, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.058, 95% CI [-0.048 to 0.164], Standard Error of Mean 0.054 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.6516, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.024, 95% CI [-0.081 to 0.130], Standard Error of Mean 0.054 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0060, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.147, 95% CI [0.042 to 0.252], Standard Error of Mean 0.053 — Olo 20 mcg qd minus Placebo

8. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-6 h (AUC 0-6h) Response at Week 4
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. FEV1 AUC 0-6h was calculated from 0-6 hours post-dose using the trapezoidal rule, divided by the observation time (6h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on first day of randomized treatment (baseline) and 30 min, 1h, 2h, 3h, 4h, 5h, 6h relative to dose at Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.091 (0.037) | 0.269 (0.035) | 0.229 (0.035) | 0.190 (0.035) | 0.323 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.178, 95% CI [0.079 to 0.277], Standard Error of Mean 0.050 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0070, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.137, 95% CI [0.038 to 0.237], Standard Error of Mean 0.051 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0512, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.099, 95% CI [-0.001 to 0.198], Standard Error of Mean 0.050 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.232, 95% CI [0.133 to 0.331], Standard Error of Mean 0.050 — Olo 20 mcg qd minus Placebo

9. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-6 h (AUC 0-6h) Response at Week 4
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to the first dose of randomized treatment. FVC AUC 0-6h was calculated from 0-6 hours post-dose using the trapezoidal rule, divided by the observation time (6h) to report in litres.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.076 (0.045) | 0.159 (0.042) | 0.154 (0.043) | 0.113 (0.043) | 0.267 (0.042)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.1811, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.082, 95% CI [-0.039 to 0.203], Standard Error of Mean 0.061 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.2118, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.077, 95% CI [-0.044 to 0.199], Standard Error of Mean 0.062 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.5504, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.037, 95% CI [-0.085 to 0.158], Standard Error of Mean 0.062 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.191, 95% CI [0.069 to 0.312], Standard Error of Mean 0.062 — Olo 20 mcg qd minus Placebo

10. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-3 h (AUC 0-3h) Response at Day 1
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. FEV1 AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on first day of randomized treatment (baseline) and 30 min, 1h, 2h, 3h relative to dose at Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.092 (0.030) | 0.271 (0.028) | 0.275 (0.028) | 0.265 (0.028) | 0.383 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.178, 95% CI [0.102 to 0.255], Standard Error of Mean 0.039 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.183, 95% CI [0.106 to 0.260], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.173, 95% CI [0.096 to 0.250], Standard Error of Mean 0.039 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.291, 95% CI [0.214 to 0.367], Standard Error of Mean 0.039 — Olo 20 mcg qd minus Placebo

11. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-3 h (AUC 0-3h) Response at Week 1
Description: as for outcome 10
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on first day of randomized treatment (baseline) and 30 min, 1h, 2h, 3h relative to dose at Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.062 (0.034) | 0.252 (0.032) | 0.258 (0.033) | 0.219 (0.032) | 0.325 (0.032)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.190, 95% CI [0.101 to 0.279], Standard Error of Mean 0.045 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.196, 95% CI [0.107 to 0.286], Standard Error of Mean 0.046 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.157, 95% CI [0.067 to 0.246], Standard Error of Mean 0.045 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.263, 95% CI [0.174 to 0.352], Standard Error of Mean 0.045 — Olo 20 mcg qd minus Placebo

12. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-3 h (AUC 0-3h) Response at Week 2
Description: as for outcome 10
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on first day of randomized treatment (baseline) and 30 min, 1h, 2h, 3h relative to dose at Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.084 (0.038) | 0.298 (0.036) | 0.240 (0.036) | 0.172 (0.036) | 0.311 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.214, 95% CI [0.115 to 0.313], Standard Error of Mean 0.050 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0021, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.156, 95% CI [0.057 to 0.255], Standard Error of Mean 0.050 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0795, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.088, 95% CI [-0.010 to 0.187], Standard Error of Mean 0.050 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.227, 95% CI [0.129 to 0.326], Standard Error of Mean 0.050 — Olo 20 mcg qd minus Placebo

13. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-3 h (AUC 0-3h) Response at Week 4
Description: as for outcome 10
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on first day of randomized treatment (baseline) and 30 min, 1h, 2h, 3h relative to dose at Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.092 (0.037) | 0.271 (0.035) | 0.224 (0.035) | 0.192 (0.035) | 0.332 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 0.179, 95% CI [0.082 to 0.276], Standard Error of Mean 0.049 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0077, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.132, 95% CI [0.035 to 0.229], Standard Error of Mean 0.049 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0427, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.100, 95% CI [0.003 to 0.197], Standard Error of Mean 0.049 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.240, 95% CI [0.143 to 0.336], Standard Error of Mean 0.049 — Olo 20 mcg qd minus Placebo

14. Secondary Outcome: Peak FEV1 (0-3h) Response At Day 1
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. Peak FEV1 (0-3h) values were obtained within 0 - 3 hours after treatment.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to 30 min, 1 h, 2 h, and 3 h relative to dose at day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.203 (0.036) | 0.372 (0.034) | 0.378 (0.034) | 0.376 (0.034) | 0.499 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.169, 95% CI [0.074 to 0.263], Standard Error of Mean 0.048 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.174, 95% CI [0.080 to 0.269], Standard Error of Mean 0.048 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.173, 95% CI [0.078 to 0.268], Standard Error of Mean 0.048 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.296, 95% CI [0.202 to 0.390], Standard Error of Mean 0.048 — Olo 20 mcg qd minus Placebo

15. Secondary Outcome: Peak FEV1 (0-3h) Response After 1 Week
Description: as for outcome 14
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to 30 min, 1 h, 2 h, and 3 h relative to dose after 1 week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.170 (0.036) | 0.343 (0.034) | 0.355 (0.034) | 0.308 (0.034) | 0.407 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.173, 95% CI [0.078 to 0.268], Standard Error of Mean 0.048 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.185, 95% CI [0.090 to 0.281], Standard Error of Mean 0.048 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0047, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.138, 95% CI [0.043 to 0.233], Standard Error of Mean 0.048 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.237, 95% CI [0.142 to 0.332], Standard Error of Mean 0.048 — Olo 20 mcg qd minus Placebo

16. Secondary Outcome: Peak FEV1 (0-3h) Response After 2 Weeks
Description: as for outcome 14
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to 30 min, 1 h, 2 h, and 3 h relative to dose after 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.182 (0.041) | 0.386 (0.039) | 0.335 (0.039) | 0.261 (0.038) | 0.403 (0.038)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.204, 95% CI [0.096 to 0.312], Standard Error of Mean 0.055 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0057, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.153, 95% CI [0.045 to 0.261], Standard Error of Mean 0.055 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1513, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.079, 95% CI [-0.029 to 0.186], Standard Error of Mean 0.055 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.221, 95% CI [0.114 to 0.328], Standard Error of Mean 0.055 — Olo 20 mcg qd minus Placebo

17. Secondary Outcome: Peak FEV1 (0-3h) Response After 4 Weeks
Description: as for outcome 14
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to 30 min, 1 h, 2 h, and 3 h relative to dose after 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.198 (0.040) | 0.363 (0.038) | 0.315 (0.038) | 0.279 (0.038) | 0.430 (0.038)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.166, 95% CI [0.060 to 0.271], Standard Error of Mean 0.054 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0307, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.117, 95% CI [0.011 to 0.223], Standard Error of Mean 0.054 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1320, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.081, 95% CI [-0.025 to 0.187], Standard Error of Mean 0.054 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.232, 95% CI [0.127 to 0.337], Standard Error of Mean 0.054 — Olo 20 mcg qd minus Placebo

18. Secondary Outcome: Peak FVC (0-3h) Response At Day 1
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FVC values prior to the first dose of randomized treatment. Peak FVC (0-3h) values were obtained within 0 - 3 hours after treatment.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to 30 min, 1 h, 2 h, and 3 h relative to dose after 1 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.218 (0.041) | 0.297 (0.039) | 0.315 (0.039) | 0.315 (0.039) | 0.398 (0.039)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.1585, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.079, 95% CI [-0.031 to 0.188], Standard Error of Mean 0.056 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0848, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.097, 95% CI [-0.013 to 0.207], Standard Error of Mean 0.056 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0838, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.097, 95% CI [-0.013 to 0.207], Standard Error of Mean 0.056 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis; Mean Difference (Final Values) = 0.180, 95% CI [0.070 to 0.289], Standard Error of Mean 0.056 — Olo 20 mcg qd minus Placebo

19. Secondary Outcome: Peak FVC (0-3h) Response After 1 Week
Description: as for outcome 18
Time Frame: as for outcome 18
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.182 (0.044) | 0.281 (0.041) | 0.301 (0.042) | 0.259 (0.042) | 0.367 (0.041)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0959, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.099, 95% CI [-0.018 to 0.216], Standard Error of Mean 0.059 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0470, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.119, 95% CI [0.002 to 0.237], Standard Error of Mean 0.060 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1960, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.077, 95% CI [-0.040 to 0.195], Standard Error of Mean 0.060 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.185, 95% CI [0.068 to 0.302], Standard Error of Mean 0.059 — Olo 20 mcg qd minus Placebo

20. Secondary Outcome: Peak FVC (0-3h) Response After 2 Weeks
Description: as for outcome 18
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.184 (0.047) | 0.327 (0.045) | 0.290 (0.045) | 0.234 (0.045) | 0.361 (0.045)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0270, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.143, 95% CI [0.016 to 0.269], Standard Error of Mean 0.064 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1031, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.106, 95% CI [-0.021 to 0.233], Standard Error of Mean 0.065 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.4378, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.050, 95% CI [-0.077 to 0.177], Standard Error of Mean 0.064 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0064, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.176, 95% CI [0.050 to 0.303], Standard Error of Mean 0.064 — Olo 20 mcg qd minus Placebo

21. Secondary Outcome: Peak FVC (0-3h) Response After 4 Weeks
Description: as for outcome 18
Time Frame: as for outcome 17
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
Liter | 0.199 (0.051) | 0.274 (0.048) | 0.267 (0.048) | 0.235 (0.048) | 0.439 (0.048)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.2781, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.075, 95% CI [-0.061 to 0.210], Standard Error of Mean 0.069 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.3284, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.068, 95% CI [-0.068 to 0.204], Standard Error of Mean 0.069 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.6020, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.036, 95% CI [-0.100 to 0.171], Standard Error of Mean 0.069 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.240, 95% CI [0.104 to 0.375], Standard Error of Mean 0.069 — Olo 20 mcg qd minus Placebo

22. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 6-12 h (AUC 6-12h) Response at Week 4
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. FEV1 AUC 6-12h was calculated from 6-12 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 hour (h) prior to dose on first day of randomized treatment (baseline) and 1h, 3h, 6h, 9h, 12h relative to dose at Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 52 | 59 | 55 | 56 | 55
Liter | 0.054 (0.051) | 0.107 (0.048) | 0.098 (0.049) | 0.092 (0.049) | 0.216 (0.049)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.4331, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.052, 95% CI 2-sided [-0.079 to 0.184], Standard Error of Mean 0.067 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.5150, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.044, 95% CI 2-sided [-0.089 to 0.178], Standard Error of Mean 0.068 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.5714, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.038, 95% CI 2-sided [-0.095 to 0.171], Standard Error of Mean 0.068 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0177, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.162, 95% CI 2-sided [0.028 to 0.296], Standard Error of Mean 0.068 — Olo 20 mcg qd minus Placebo

23. Secondary Outcome: Weekly Mean Evening PEFR After 4 Weeks
Description: Response was defined as change from baseline. Baseline PEFR was defined as the mean of the evening PEFR measurements obtained during the week just prior to first dose of randomized treatment.
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter/minute
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 59 | 61
Liter/minute | 384.08 (5.585) | 407.05 (5.256) | 408.68 (5.297) | 420.88 (5.341) | 426.58 (5.258)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0030, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 22.970, 95% CI 2-sided [7.883 to 38.057], Standard Error of Mean 7.665 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 24.600, 95% CI 2-sided [9.446 to 39.754], Standard Error of Mean 7.700 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 36.806, 95% CI 2-sided [21.598 to 52.015], Standard Error of Mean 7.727 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 42.505, 95% CI 2-sided [27.399 to 57.611], Standard Error of Mean 7.675 — Olo 20 mcg qd minus Placebo

24. Secondary Outcome: PEFR Variability After 4 Weeks
Description: PEFR variability represents the absolute difference between the highest morning PEFR value and the highest evening PEFR value of 1 day, divided by the arithmetic mean of these 2 PEFR values and expressed as a percent, weekly means.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of PEFR
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 59 | 61
percentage of PEFR | 11.694 (0.780) | 10.575 (0.736) | 9.343 (0.739) | 8.649 (0.747) | 8.756 (0.733)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.2898, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.118, 95% CI 2-sided [-3.194 to 0.957], Standard Error of Mean 1.055 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0270, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.351, 95% CI 2-sided [-4.432 to -0.269], Standard Error of Mean 1.057 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0045, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.045, 95% CI 2-sided [-5.138 to -0.952], Standard Error of Mean 1.063 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0056, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.937, 95% CI 2-sided [-5.010 to -0.865], Standard Error of Mean 1.053 — Olo 20 mcg qd minus Placebo

25. Secondary Outcome: Weekly Mean Number of Occasions of Rescue Therapy After 4 Weeks
Description: Weekly mean number of occasions of rescue therapy used per day (prn salbutamol [albuterol]) as assessed by the e-Diary (e-Diary incorporated in AM2+).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of Puffs
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 59 | 61
Number of Puffs | 1.449 (0.190) | 1.162 (0.179) | 0.923 (0.181) | 1.117 (0.182) | 0.856 (0.179)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.2645, ANCOVA; Analysis of covariance model with terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = -0.287, 95% CI 2-sided [-0.793 to 0.218], Standard Error of Mean 0.257 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0423, ANCOVA; Analysis of covariance model with terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = -0.526, 95% CI 2-sided [-1.034 to -0.018], Standard Error of Mean 0.258 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.2008, ANCOVA; Analysis of covariance model with terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = -0.332, 95% CI 2-sided [-0.842 to 0.178], Standard Error of Mean 0.259 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0218, ANCOVA; Analysis of covariance model with terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = -0.593, 95% CI 2-sided [-1.098 to -0.087], Standard Error of Mean 0.257 — Olo 20 mcg qd minus Placebo

26. Secondary Outcome: Area Under Curve From 0 to 3 Hours (AUC0-3)
Description: AUC0-3 represents the area under the concentration curve of olodaterol and olodaterol glucuronide (a metabolite of olodaterol) in plasma from 0 to time t=3
Time Frame: 30 minutes (mins) before drug administration and 5mins, 10mins, 20mins, 40mins, 1 hour (h) and 3h after drug administration
Population: All evaluable patients were included in the pharmacokinetic (PK) analysis. A patient was considered to be not evaluable if the patient had a protocol violation relevant to the evaluation of PK parameters or had insufficient data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hours/milliliter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 0 | 28 | 44
Picogram*hours/milliliter
  Olodaterol (N=0;0;0;20;44) |  |  |  | 11.8 (35.2) | 17.8 (42.1)
  Olodaterol glucuronide (N=0;0;0;28;36) |  |  |  | 9.14 (48.6) | 20.3 (48.0)

27. Secondary Outcome: Maximum Concentration (Cmax)
Description: Cmax represents the maximum concentration of olodaterol and olodaterol glucuronide (a metabolite of olodaterol) in plasma.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram/milliliter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 38 | 54 | 58
Picogram/milliliter
  Olodaterol (N=0;0;21;44;58) |  |  | 3.54 (48.4) | 4.63 (59.7) | 8.24 (68.6)
  Olodaterol glucuronide (N=0;0;38;54;57) |  |  | 3.57 (82.1) | 5.00 (50.4) | 9.54 (69.7)

28. Secondary Outcome: Time From Dosing to the Maximum Concentration (Tmax)
Description: tmax represents the time from dosing to maximum concentration of olodaterol and olodaterol glucuronide (a metabolite of olodaterol) in plasma.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 38 | 54 | 58
hours
  Olodaterol (N=0;0;21;44;58) |  |  | 0.183 [0.0830 to 2.97] | 0.234 [0.0830 to 2.83] | 0.267 [0.0670 to 1.07]
  Olodaterol glucuronide (N=0;0;38;54;57) |  |  | 2.97 [0.117 to 3.05] | 2.97 [0.233 to 3.20] | 2.97 [0.100 to 3.22]

29. Secondary Outcome: Area Under Curve From 0 to 3 Hours at Steady State (AUC0-3,ss)
Description: AUC0-3,ss represents the area under the concentration curve of olodaterol and olodaterol glucuronide (a metabolite of olodaterol) in plasma from 0 to time t=3 at steady state.
Time Frame: 30 minutes (mins) before drug administration and 5mins, 10mins, 20mins, 40mins, 1 hour (h), 3h and 6h after drug administration
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hours/milliliter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 38 | 44 | 54
Picogram*hours/milliliter
  Olodaterol (N=0;0;0;38;53) |  |  | NA (NA) — No patients analyzed. | 13.0 (42.7) | 25.5 (56.5)
  Olodaterol glucuronide (N=0;0;38;44;54) |  |  | 7.71 (62.2) | 9.04 (64.2) | 19.0 (59.4)

30. Secondary Outcome: Area Under Curve From 0 to 6 Hours at Steady State (AUC0-6,ss)
Description: AUC0-6,ss represents the area under the concentration curve of olodaterol and olodaterol glucuronide (a metabolite of olodaterol) in plasma from 0 to time t=6 at steady state.
Time Frame: as for outcome 29
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hours/milliliter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 21 | 32 | 50
Picogram*hours/milliliter
  Olodaterol (N=0;0;0;32;50) |  |  | NA (NA) — No patients analyzed. | 25.3 (35.7) | 46.3 (50.3)
  Olodaterol glucuronide (N=0;0;21;23;33) |  |  | 19.2 (58.2) | 21.3 (56.4) | 37.6 (54.2)

31. Secondary Outcome: Area Under Curve From 0 to 24 Hours at Steady State (AUC0-24,ss)
Description: AUC0-24,ss represents the area under the concentration curve of olodaterol and olodaterol glucuronide (a metabolite of olodaterol) in plasma from 0 to time t=24 at steady state.
Time Frame: as for outcome 29
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hours/milliliter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 0 | 20 | 44
Picogram*hours/milliliter
  Olodaterol |  |  |  | 83.7 (30.3) | 147 (49.5)
  Olodaterol glucuronide |  |  |  | NA (NA) — No patients analyzed. | NA (NA) — No patients analyzed.

32. Secondary Outcome: Maximum Concentration at Steady State (Cmax,ss)
Description: Cmax,ss represents the maximum concentration of olodaterol and olodaterol glucuronide (a metabolite of olodaterol) in plasma at steady state.
Time Frame: as for outcome 29
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram/milliliter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 46 | 46 | 56
Picogram/milliliter
  Olodaterol N=(0;0;39;45;56) |  |  | 3.19 (35.0) | 5.09 (53.0) | 12.1 (69.2)
  Olodaterol glucuronide N=(0;0;46;46;54) |  |  | 4.16 (46.8) | 5.04 (57.4) | 9.19 (53.6)

33. Secondary Outcome: Time From Dosing to the Maximum Concentration at Steady State (Tmax,ss)
Description: tmax,ss represents the time from dosing to maximum concentration of olodaterol and olodaterol glucuronide (a metabolite of olodaterol) in plasma at steady state.
Time Frame: as for outcome 29
Population: as for outcome 26
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 46 | 46 | 56
hours
  Olodaterol (N=0;0;39;45;56) |  |  | 0.333 [0.0830 to 2.92] | 0.333 [0.0830 to 2.93] | 0.333 [0.0830 to 1.08]
  Olodaterol glucuronide (N=0;0;46;46;54) |  |  | 3.00 [0.100 to 6.00] | 3.00 [0.917 to 6.02] | 2.97 [0.350 to 6.05]

34. Secondary Outcome: Total Score in Asthma Control Questionnaire After 4 Weeks
Description: Adequacy of asthma control was assessed using a scale of: 0=totally controlled, to 6=Severely uncontrolled.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 53 | 58 | 58 | 59 | 60
units on a scale | 1.456 (0.089) | 1.314 (0.086) | 1.260 (0.086) | 1.129 (0.084) | 1.181 (0.084)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.2156, ANCOVA; Analysis of covariance model with terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = -0.142, 95% CI [-0.368 to 0.083], Standard Error of Mean 0.114 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0869, ANCOVA; Analysis of covariance model with terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = -0.197, 95% CI [-0.422 to 0.029], Standard Error of Mean 0.114 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0044, ANCOVA; Analysis of covariance model with terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = -0.328, 95% CI [-0.552 to -0.103], Standard Error of Mean 0.114 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0158, ANCOVA; Analysis of covariance model with terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = -0.276, 95% CI [-0.499 to -0.052], Standard Error of Mean 0.113 — Olo 20 mcg qd minus Placebo

35. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, ECG and Physical Examination
Description: Clinical relevant abnormalities for vital signs, ECG and physical examination. Any new or clinically relevant worsening of baseline conditions was reported as adverse events.
Time Frame: 4 weeks
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 54 | 61 | 60 | 60 | 61
participants
  Palpitations | 0 | 0 | 1 | 0 | 2
  Ventricular extrasystoles | 0 | 0 | 1 | 0 | 0
  Blood creatine phosphokinase increased | 0 | 0 | 0 | 0 | 1

36. Secondary Outcome: Laboratory Testing: Average Change From Baseline of Potassium
Description: Laboratory testing: Average change from baseline of potassium measured on test-days. Pre-dose value on test day 1 is the baseline value.
Time Frame: Baseline and 29 days
Population: Treated Set
Measure: Geometric Mean (Inter-Quartile Range); unit: mmol/L
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 51 | 54 | 52 | 56 | 57
mmol/L | 0.98 (NA) [0.94 to 1.02] | 0.97 (NA) [0.93 to 1.02] | 1.00 (NA) [0.95 to 1.05] | 0.99 (NA) [0.96 to 1.03] | 0.97 (NA) [0.92 to 1.02]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/61 | 0/60 | 1/60 | 1/61
Other Adverse Events (participants affected / at risk) | 9/54 | 9/61 | 11/60 | 7/60 | 11/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | Olo 2 mcg qd (N=61) | Olo 5 mcg qd (N=60) | Olo 10 mcg qd (N=60) | Olo 20 mcg qd (N=61)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | Olo 2 mcg qd (N=61) | Olo 5 mcg qd (N=60) | Olo 10 mcg qd (N=60) | Olo 20 mcg qd (N=61)
Nasopharyngitis (Infections and infestations) | 4 | 4 | 5 | 3 | 2
Headache (Nervous system disorders) | 3 | 4 | 4 | 3 | 5
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication